CLINICAL TRIAL: NCT04937179
Title: The Effect of Ischemic Conditioning on Strength and Ambulation in Subjects with Peripheral Artery Disease (PAD)
Brief Title: The Effect of Ischemic Conditioning on Strength and Ambulation in Subjects with PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Lindsay Hannigan, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021-0223; 20CDA35310419 (Other: American Heart Association)
Record Dates: First submitted 2021-05-27; First posted 2021-06-23 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Disease; Amputation; Lower Limb Amputation Knee; Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation Below Knee (Injury)
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ischemic Conditioning Low (Sham Comparator): Blood flow restriction with low compression
  Interventions: Procedure: Ischemic Conditioning Low - Sham Comparator
- Ischemic Conditioning High (Active Comparator): Blood flow restriction with high compression
  Interventions: Procedure: Ischemic Conditioning High - Active Comparator

INTERVENTIONS:
Procedure: Ischemic Conditioning Low - Sham Comparator — The use of a Hokanson rapid inflator cuff to restrict blood flow at 25mmHg for 5 minutes followed by a 5 minute reperfusion period, repeated for 5 cycles.
  Arms: Ischemic Conditioning Low
Procedure: Ischemic Conditioning High - Active Comparator — The use of a Hokanson rapid inflator cuff to restrict blood flow at 225mmHg for 5 minutes followed by a 5 minute reperfusion period, repeated for 5 cycles.
  Arms: Ischemic Conditioning High

SUMMARY:
Lower limb amputation is common in the United States, with approximately 150,000 amputations annually. Most individuals walking with a prosthesis demonstrate asymmetrical loading-i.e., they favor the amputated side by placing more weight and increased ground reaction forces through the intact limb-which likely contributes to increased metabolic cost of walking. Lack of adequate muscular strength in the lower limb to attenuate these forces places increased stress on the joints, which may be displaced proximally, and may play a role in reported knee and hip pain in the intact limb.

Lower limb muscle weakness following amputation has been well documented. Increasing quadriceps strength is important after an amputation because it is positively correlated with gait speed. Gait speed may also be associated with successful community mobility, which leads to improved quality of life following amputation. Individuals with amputation who resume an active lifestyle are able to maintain strength. However, these individuals represent a minority of persons with lower limb amputation; most individuals report more barriers than motivators to adopt an active lifestyle.

Ischemic conditioning (IC) may strengthen leg muscles and reduce the metabolic cost of activity after amputation. In IC, the limb is exposed to brief, repeated bouts of ischemia (reduced blood flow) immediately followed by reperfusion. IC has been shown to improve muscle performance in healthy and diseased populations. IC has also been used more recently in patients with peripheral artery disease (PAD) as an intervention to improve function, such as walking ability. Acute exposure to IC increases muscle strength and activation, both in healthy, active individuals and in those with severe neuromuscular dysfunction, such as stroke survivors. IC also attenuates muscular fatigue. Increased fatigue resistance at submaximal contraction levels following IC may be due to increased neural activation of skeletal muscle. Changes in neural activation of muscle may be particularly beneficial during cortical reorganization after amputation. Reduced quadriceps fatigue during submaximal activities may also drive changes in gait kinematics, such as increased knee flexion during loading and mid-stance. Exposure to IC may also increase the oxidative properties of skeletal muscle, offering a direct pathway to reduce metabolic cost. Therefore, IC may lead to cellular changes that lower the metabolic cost of activity.

The primary aim of this study is to quantify the benefits of acute and chronic IC on quadriceps strength and walking economy in individuals with PAD and history of lower limb amputation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Able to ambulate independently without the use of aids (i.e., walking cane)
* Able to walk at least 10 minutes continuously without stopping
* History of diagnosed peripheral artery disease.
* For Amputees: History lower limb unilateral transtibial or transfemoral amputation.

Exclusion Criteria:

* Inability to give informed consent
* neurological disorder that affects gait
* two or more falls within the previous 12 months
* currently pregnant (or intend to become pregnant while participating in study)
* history of any condition where fatiguing contractions or resisted leg contractions are contraindicated
* blood clots in the leg, or any condition in which compression of the thigh or transient ischemia is contraindicated (e.g. open wounds in the leg).
* history of hypertension
* history of heart failure
* Head injury within the previous 6 months
* Seizure disorder
* Adverse reaction to ultrasound gel
* History of thrombosis
* History of sickle cell trait

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in quadriceps strength | through study completion, an average of 6 weeks
  Quadriceps strength assessed by a Biodex dynamometer
Change in gait kinematics | through study completion, an average of 6 weeks
  Gait mechanics assessed by joint angles using Vicon cameras and reflective markers
Change in gait kinetics | through study completion, an average of 6 weeks
  Gait mechanics assessed by joint forces using a Bertec instrumented treadmill in combination with gait kinematics
Change in gait metabolics | through study completion, an average of 6 weeks
  Assessment of oxygen consumption during walking using a metabolic cart

SECONDARY OUTCOMES:
Six-minute walk test | through study completion, an average of 6 weeks
  Measurement of distance walked in six minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Slater, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- UIC Physical Therapy Faculty Practice, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No